CLINICAL TRIAL: NCT03579342
Title: Using App-technology and a Personalized Health Plan to Improve Lifestyle Habits Among Working Adults - a Randomized Controlled Trial
Brief Title: App-technology to Improve Healthy Lifestyle Behaviors Among Working Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Research Institutes of Sweden (Other)
Responsible Party: Principal Investigator, Ylva Trolle Lagerros, MD, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/411-31
Record Dates: First submitted 2018-05-08; First posted 2018-07-06 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Lifestyle; Quality of Life; mHealth; Mobile Applications; Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App technology and coaching (Experimental): Participants in the intervention group with app technology and coaching participate in a first meeting with the coach and will thereafter receive active support from the coach every 4 weeks for the duration of the intervention.
  Interventions: Behavioral: App-technology and active coaching to improve lifestyles behaviors
- App technology only (Experimental): Participants in the intervention group with only app technology participate in a first meeting with the coach but do not get any additional support during follow-up.
  Interventions: Behavioral: App-technology to improve lifestyle behaviors
- Control group (No Intervention): Participants in the control group participate in baseline assessments. The control group will get access to the app and will have a meeting with a coach after 12 weeks of follow-up.

INTERVENTIONS:
Behavioral: App-technology and active coaching to improve lifestyles behaviors — Access to the smartphone-app during 12 weeks. A personal health goal related to for example diet, physical activity or stress habits, is set together with a heath coach. Participants receive continuous coaching every 4 weeks during follow-up.
  Arms: App technology and coaching
Behavioral: App-technology to improve lifestyle behaviors — Access to the smartphone-app during 12 weeks. A personal health goal related to for example diet, physical activity or stress habits, is set together with a heath coach. Participants receive continuous coaching every 4 weeks during follow-up.
  Arms: App technology only

SUMMARY:
The aim of this study is to evaluate if modern technology such as smartphone applications can be used to facilitate lifestyle changes and thereby improve health-related quality of life in gainfully employed persons in the general population in Stockholm, Sweden. The hypothesis is that at follow-up, the intervention group that use the new application will have improved health-related quality of life and other lifestyle habits including diet, physical activity and sleep, as well as biomarkers, compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to communicate in Swedish
* Have access to and use a smartphone

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Health related quality of life assessed by the RAND-36 questionnaire | 12-weeks follow-up
  Mental and Physical Health Scores (range 0-100) are assessed using 36 questions

SECONDARY OUTCOMES:
Physical activity | Baseline (week 0) and at 12-weeks follow-up
  Minutes per day spent on a sedentary, light, moderate or higher activity level assessed using accelerometers
HbA1c (Heamoglobin A1c) | Baseline (week 0) and at 12-weeks follow-up
  mmol/mol
Total cholesterol | Baseline (week 0) and at 12-weeks follow-up
  (mmol/L)
Apolipoprotein A1 | Baseline (week 0) and at 12-weeks follow-up
  (g/l)
Apolipoprotein B | Baseline (week 0) and at 12-weeks follow-up
  (g/l)
Body Mass Index | Baseline (week 0) and at 12-weeks follow-up
  (kg/m2)
Body weight | Baseline (week 0) and at 12-weeks follow-up
  (kg)
Waist circumference | Baseline (week 0) and at 12-weeks follow-up
  (cm)
Body composition | Baseline (week 0) and at 12-weeks follow-up
  (%Body Fat)
Blood pressure (Systolic and Diastolic) | Baseline (week 0) and at 12-weeks follow-up
  (mmHg)

OTHER OUTCOMES:
Change in dietary habits | Baseline (week 0) and at 12-weeks follow-up
  Intake of macro- and Micro nutrients are assessed based on responses to a food frequency questionnaire
Change in eating behaviors according to the Three Factor Eating Questionnaire (TFEQ) | Baseline (week 0) and at 12-weeks follow-up
  Emotional eating, uncontrolled eating, and cognitive restricted eating are assessed using a 21-item questionnaire
Change in tobacco use (user/non-user) | Baseline (week 0) and at 12-weeks follow-up
  Smoking and Swedish snuff use
Change in sleeping habits | Baseline (week 0) and at 12-weeks follow-up
  Assessed using a modified 13-item Karolinska Sleep questionnaire
Change in perceived Purpose In Life (PIL) | Baseline (week 0) and at 12-weeks follow-up
  6-item questionnaire
Change in perceived stress levels | Baseline (week 0) and at 12-weeks follow-up
  Assessed using the 14-item perceived stress scale (PSS)
Change in motivation to make lifestyle changes | Baseline (week 0) and at 12-weeks follow-up
  Assessed using Prochaskas' transtheoretical model of behavior change
Social support for an overall healthy lifestyle | Baseline (week 0)
  Social support for maintenance of a healthy Lifestyle from family, friends and co-workers is assessed by a 5-item questionnaire
Change in self-reported sitting time and physical activity | Baseline (week 0) and at 12-weeks follow-up
  Assessed by 6 questions on sitting time and exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Select One..., Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonn S, Licitra G, Bellocco R, Trolle Lagerros Y. Clinical Outcomes Among Working Adults Using the Health Integrator Smartphone App: Analyses of Prespecified Secondary Outcomes in a Randomized Controlled Trial. J Med Internet Res. 2022 Mar 21;24(3):e24725. doi: 10.2196/24725. PMID 35311677
- [Derived] Melin J, Bonn SE, Pendrill L, Trolle Lagerros Y. A Questionnaire for Assessing User Satisfaction With Mobile Health Apps: Development Using Rasch Measurement Theory. JMIR Mhealth Uhealth. 2020 May 26;8(5):e15909. doi: 10.2196/15909. PMID 32452817
- [Derived] Bonn SE, Lof M, Ostenson CG, Trolle Lagerros Y. App-technology to improve lifestyle behaviors among working adults - the Health Integrator study, a randomized controlled trial. BMC Public Health. 2019 Mar 7;19(1):273. doi: 10.1186/s12889-019-6595-6. PMID 30845949